CLINICAL TRIAL: NCT04970654
Title: A Trial Comparing the Efficacy and Safety of Once Weekly Dosing of Somapacitan With Daily Norditropin® in Chinese Children With Growth Hormone Deficiency
Brief Title: A Research Study in Chinese Children With a Low Level of Hormone to Grow. Treatment is Somapacitan Once a Week Compared to Norditropin® Once a Day.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4468; U1111-1250-7530 (Other: World Health Organization); 2020-002974-28 (Other: European Medicines Agency (EudraCT))
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Growth Hormone Deficiency in Children
MeSH Terms: interventions — somapacitan; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Somapacitan weekly (Experimental): participants will receive once-weekly somapacitan for 52 weeks
  Interventions: Drug: somapacitan
- Norditropin® daily (Active Comparator): Participants will receive Norditropin® daily for 52 weeks
  Interventions: Drug: Norditropin®

INTERVENTIONS:
Drug: somapacitan — Somapacitan (0.16 mg/kg/week) will be administered subcutaneously (s.c.; under the skin) once weekly by PDS290 pen-injector. Somapacitan can be injected any time during the once weekly dosing day. The dose will be calculated based on the subject's current body weight.
  Arms: Somapacitan weekly
Drug: Norditropin® — Norditropin® (0.034 mg/kg/day) will be administered s.c. once daily by FlexPro® pen-injector. Norditropin® should be injected daily in the evening. The dose will be calculated based on the subject's current body weight.
  Arms: Norditropin® daily

SUMMARY:
The study compares two medicines for children with a low level of hormone to grow: somapacitan (a new medicine) given once a week and Norditropin® (a medicine doctors can already prescribe) given once a day. Researchers will test somapacitan to see how well it works, compared to the standard treatment with Norditropin®. The participants will either get Norditropin® once every day or somapacitan once every week - which treatment the participant gets is decided by chance. The participant and the study doctor will know which treatment the participant gets. The study includes a 52 week treatment period and a minimum of 30 days follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent or legally acceptable representative of participant and child assent, as age-appropriate must be obtained before any trial related activities
* The parent or legally acceptable representative of the child must sign and date the Informed consent form (according to local requirements)
* The child must sign and date child assent form or provide oral assent (if required according to local requirements)
* Prepubertal children: a) Boys: Age more than or equal to 2 years and 26 weeks and less than or equal to 11.0 years at the time of signing informed consent.
* Testis volume less than 4 ml. b) Girls: Age more than or equal to 2 years and 26 weeks and less than or equal to 10.0 years at the time of signing informed consent. Tanner stage 1 for breast development (no palpable glandular breast tissue)
* Confirmed diagnosis of growth hormone deficiency determined by two different growth hormone stimulation tests performed within 12 months prior to randomisation, defined as a peak growth hormone level of less than or equal to 10.0 ng/ml using the WHO International Somatropin 98/574 standard
* If only one growth hormone stimulation test is available before screening, then confirmation of growth hormone deficiency by second and different growth hormone stimulation test must be done
* For children with at least 2 additional pituitary hormone deficiencies (other than growth hormone deficiency) only one growth hormone stimulation test is needed
* Impaired height defined as at least 2.0 standard deviations below the mean height for chronological age and gender according to Chinese general population standards at screening
* Impaired height velocity defined as annualised height velocity at screening less than 7cm/year for subjects between 2.5 and 3 years old and less than 5 cm/year for subjects from 3 years and above calculated over a time span of minimum 3 months and maximum 18 months prior to screening according to Chinese guideline and expert consensus on children with short stature and GH therapy
* No prior exposure to growth hormone therapy or IGF-I treatment
* Bone age less than chronological age at screening
* Body Mass Index more than 5th and less than 95th percentile, Body Mass Index-for-age growth charts according to Chinese general population standards.
* IGF-I < -1.0 SDS at screening, compared to age and gender normalized range measured at central laboratory
* No intracranial tumour confirmed by magnetic resonance imaging or computer tomography scan. An image or scan taken within 9 months prior to screening can be used as screening data if the medical evaluation and conclusion is available

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Previous participation in this trial. Participation is defined as randomisation.
* Receipt of any investigational medicinal product within 3 months before screening or participation in another clinical trial before randomisation
* Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with standing height measurements:
* Turner Syndrome (including mosaicisms)
* Chromosomal aneuploidy and significant gene mutations causing medical "syndromes" with short stature, including but not limited to Laron syndrome, Noonan syndrome, Prader-Willi Syndrome, abnormal SHOX-1 gene analysis or absence of GH receptors
* Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants
* Congenital abnormalities (causing skeletal abnormalities), including but not limited to Russell-Silver Syndrome or skeletal dysplasias
* Family history of skeletal dysplasia
* Children born small for gestational age (birth weight 10th percentile of the recommended gender-specific birth weight for gestational age according to national standards in China5
* Children diagnosed with diabetes mellitus or screening values from central laboratory of

  1. fasting plasma glucose more than or equal to 126 mg/dl (7.0 mmol/L) or
  2. HbA1c more than or equal to 6.5 %
* Current inflammatory diseases requiring systemic corticosteroid treatment for longer than 2 consecutive weeks within the last 3 months prior to screening
* Children requiring inhaled glucocorticoid therapy at a dose greater than 400 µg/day of inhaled budesonide or equivalents for longer than 4 consecutive weeks within the last 12 months prior to screening
* Concomitant administration of other treatments that may have an effect on growth, e.g. but not limited to methylphenidate for treatment of attention deficit hyperactivity disorder (ADHD)
* Diagnosis of attention deficit hyperactivity disorder
* Prior history or presence of malignancy including intracranial tumours
* Prior history or known presence of active Hepatitis B or Hepatitis C (exceptions to this exclusion criterion is the presence of antibodies due to vaccination against Hepatitis B)
* Any clinically significant abnormal laboratory screening tests, as judged by the study doctor
* Any disorder which, in the opinion of the study doctor, might jeopardise Participant's safety or compliance with the protocol
* The participant or the parent/legally acceptable representative is likely to be non-compliant in respect to trial conduct, as judged by the study doctor
* Children with hypothyroidism and/or adrenal insufficiency not on adequate and stable replacement therapy for at least 90 days prior to randomisation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (32):
- China (32):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Capital Center for Children's Health, Capital Medical University-Endocrinology, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University-Pediatric, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University-Pediatric, Guangzhou, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital-Endocrine Genetics and Metabolism, Zhengzhou, Henan
  - Henan Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST-Pediatric, Wuhan, Hubei
  - Hunan Children's Hospital-Child Health Center, Changsha, Hunan
  - Hunan Children's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Shaoyang University-Pediatric, Shaoyang, Hunan
  - Jiangxi Provincial Children's Hospital-Endocrine Genetics and Metabolism, Nanchang, Jiangsu
  - Children's Hospital of Soochow University-Endocrine Genetics and Metabolism, Suzhou, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Children's Hospital-Pediatric Endocrinology, Wuxi, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - The First Hospital of Jiaxing-Pediatric, Jiaxing, Jiangxi
  - The First Hospital of Jiaxing, Jiaxing, Jiangxi
  - Pingxiang Maternal and Child Health Care Hospital-Child Health Care, Pingxiang, Jiangxi
  - Pingxiang Maternal and Child Health Care Hospital, Pingxiang, Jiangxi
  - The First Bethune Hospital of Jilin University-Pediatric, Changchun, Jilin
  - The First Bethune hospital of Jilin University-Endocrinology, Changchun, Julin
  - Shandong Provincial Hospital-Pediatric, Jinan, Shandong
  - Women & Children's Health Care Hospital of Linyi-Endocrine Genetics and Metabolism, Linyi, Shandong
  - Qingdao Women and Children's Hospital-Pediatric Endocrinology&Metabolism, Qingdao, Shandong
  - Qingdao Women and Children's Hospital, Qingdao, Shandong
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Wuhan Children Hospital-Endocrine Genetics and Metabolism, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 20 sites in China.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive either somapacitan or Norditropin.
Groups:
- Norditropin: Participants received Norditropin 0.034 mg/kg (milligram per kilogram) subcutaneous injection once daily using PDS290 pen injector for 52 weeks.
- Somapacitan: Participants received somapacitan 0.16 mg/kg subcutaneous injection once weekly using PDS290 pen injector for 52 weeks.
Period: Overall Study
Arm/Group | Norditropin | Somapacitan
Started | 36 | 74
Full Analysis Set | 36 | 74
Safety Analysis Set | 36 | 74
Completed | 32 | 71
Not Completed | 4 | 3
Not completed — Withdrawal by parents/guardian | 1 | 2
Not completed — Unclassified | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Norditropin | Somapacitan | Total
Number analyzed (Participants) | 36 | 74 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.5 (2.3) | 6.6 (2.1) | 6.5 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 30 | 65 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 74 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity
Description: Height velocity (HV) was derived from height measurements taken at baseline (week 0) and the week 52 visit as: HV = (height at 52 weeks visit - height at baseline)/(time from baseline to 52 weeks visit in years).
Time Frame: Baseline (Week 0); Week 52
Population: FAS included all randomized participants. Here, Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Cm/year (centimeter per year)
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 71
Cm/year (centimeter per year) | 10.5 (2.3) | 11.0 (2.1)
Statistical Analysis 1: Comparison: Norditropin vs Somapacitan; Hypothetical strategy estimand. Height velocity at 52 weeks was analyzed using a mixed model for repeated measurements, with treatment, gender, age group, growth hormone (GH) peak group and gender by age group interaction term as factors and baseline height as a covariate, all nested within week as a factor; Test type: Non-Inferiority — Non-inferiority was considered confirmed if the lower bound of the 95% confidence interval was higher than the margin of -2.0 cm/year; Treatment difference = 0.6, 95% CI 2-sided [-0.2 to 1.3]

2. Secondary Outcome: Change in Bone Age
Description: Change in bone age is presented from week -2 to week 52. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Week -2, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 68
Years | 5.6 (2.2) | 5.5 (2.1)

3. Secondary Outcome: Change in Height Standard Deviation Score
Description: Change in the height standard deviation score (HSDS) is presented from baseline (week 0) to week 52. HSDS was derived using Chinese general population standards. The formula to calculate HSDS is: HSDS = ((Height / M)**L-1) / (L*S). L: The sex and age-specific power in the Box-Cox transformation, M: The sex and age-specific median, S: The sex and age-specific generalized coefficient of variation. The range for HSDS was -10 to +10. Negative scores indicated a height below the mean height for a child with the same age and gender, whereas positive scores indicated a height above the mean height for a child with the same age and gender. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 69
Score on a scale | 1.13 (0.48) | 1.21 (0.46)

4. Secondary Outcome: Change in Height Velocity Standard Deviation Score
Description: Change in height velocity standard deviation score (HVSDS) is presented from baseline (week 0) to week 52. HVSDS was derived using Prader standards. HVSDS was calculated using the formula: HVSDS = (height velocity - mean)/standard deviation (SD), where height velocity was the height velocity variable measured, mean and SD of height velocity by gender and age for the reference population. The range for HVSDS was -10 to +10. Negative scores indicated a height velocity below the mean height velocity for a child with the same age and gender, whereas positive scores indicated a height velocity above the mean height velocity for a child with the same age and gender. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 69
Score on a scale | 8.34 (3.01) | 8.96 (3.53)

5. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose is presented from baseline (week 0) to week 52. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: Safety analysis set (SAS): SAS included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product. Here, Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/l (milimoles per liter)
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 68
mmol/l (milimoles per liter) | 0.541 (0.523) | 0.304 (0.521)

6. Secondary Outcome: Change in HbA1c
Description: Change in glycosylated haemoglobin (HbA1c) is presented from baseline (week 0) to week 52 is presented. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: SAS included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product. Here, Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 69
Percentage (%) of HbA1c | 0.09 (0.31) | 0.19 (0.25)

7. Secondary Outcome: Change in IGF-I Standard Deviation Score
Description: Change in Insulin like growth factor-I (IGF-I) standard deviation score is presented from baseline (week 0) to week 52. The range for IGF-I SDS was from -10 to +10. Negative scores indicated a IGF-I below the mean IGF-I for a child with the same age and gender, whereas positive scores indicated a IGF-I above the mean IGF-I for a child with the same age and gender. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 67
Score on a scale | 1.73 (1.00) | 2.09 (1.28)

8. Secondary Outcome: Change in IGFBP-3 Standard Deviation Score
Description: Change in Insulin like growth factor binding protein 3 (IGFBP-3) standard deviation score is presented from baseline (week 0) to week 52. The range for IGFBP-3 SDS was from -10 to +10. Negative scores indicated a IGFBP-3 below the mean IGFBP-3 for a child with the same age and gender, whereas positive scores indicated a IGFBP-3 above the mean IGFBP-3 for a child with the same age and gender. This outcome measure was analysed based on the 'on treatment' observation period. On treatment observation period: It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 32 | 67
Score on a scale | 0.93 (0.75) | 1.06 (0.87)

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to week 57
Description: All presented AEs are TEAEs (treatment emergent adverse events). AEs with onset during the on-treatment observation period (It starts from first administration of trial product and up until last trial contact, visit 7 (52 weeks+5 days) or 14 days after last administration, whichever comes first) were considered treatment-emergent. Results are based on the SAS which included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Arm/Group | Norditropin | Somapacitan
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/36 | 8/74
Other Adverse Events (participants affected / at risk) | 29/36 | 60/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (N=36) | Somapacitan (N=74)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (N=36) | Somapacitan (N=74)
Blood glucose increased (Investigations) | 2 (2) | 2 (3)
Bronchitis (Infections and infestations) | 4 (8) | 7 (7)
COVID-19 (Infections and infestations) | 7 (7) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 12 (22)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 3 (3)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 18 (23)
Respiratory tract infection (Infections and infestations) | 5 (9) | 9 (17)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 15 (24) | 40 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04970654/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT04970654/SAP_001.pdf